CLINICAL TRIAL: NCT01651156
Title: Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel Phase 3 Study to Evaluate the Efficacy and Safety of Tolvaptan in the Treatment of Patients With Cardiac Edema Based on the Conventional Therapy
Brief Title: Efficacy and Safety Study of Tolvaptan to Treat Patients With Cardiac Edema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-12-809-01
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Cardiac Edema
MeSH Terms: conditions — Edema, Cardiac | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Frequency: once per day Duration: 7days
  Interventions: Drug: Placebo
- Tolvaptan (Experimental): Tolvaptan tablet Frequency: once per day Duration: 7days
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — oral taken
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Placebo
  Arms: placebo

SUMMARY:
A randomized, double-blind, multicenter, placebo-controlled, parallel study to evaluate the efficacy and safety of Tolvaptan in the treatment of patients with cardiac edema (body fluid retention caused by congestive heart failure) based on the conventional therapy.

To evaluate the efficacy and safety of Tolvaptan 15 mg on congestive heart failure patients with body fluid retention after current diuretic treatment, after continuous treatment of 7 days' oral Tolvaptan 15mg or placebo.

DETAILED DESCRIPTION:
* A randomized, double-blind, multicenter, placebo-controlled, parallel study
* Study population: The congestive heart failure patients with body fluid retention after received current diuretics therapy
* Number of patients: Patients will be randomly assigned to Tolvaptan and placebo group in 1:1 ratio, 120 patients in each group, 240 patients in total
* Group assignment method: Tolvaptan 15 mg group: conventional therapy + Tolvaptan 15 mg Placebo group: conventional therapy + placebo
* Administration and dosage of the study drug: Once daily, 1 tablet be taken orally after breakfast, for successive 7 days
* Study period:
* Screening period (4 days in minimum, 7 days in maximum), including:

Screening period: from the time the informed consent form is signed to Day -4 Observation period: 3 days before drug administration

* Treatment period: 7 days
* Follow up visits: Day 8 (efficacy evaluation day) and Day 7 (+3) after the last dosing
* Post treatment survey: Day 14 (+3) after the last dosing

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with one of the oral diuretic therapy standards （include the patients who will be treated with one of the oral diuretic therapy standards from the beginning of the observation period）:

  1. Only 40 mg/day furosemide taken orally or other oral loop diuretics equivalent to 40 mg/day furosemide note 1)
  2. Combination treatment of oral loop diuretics and thiazide diuretics (no dosage limitation)
  3. Combination treatment of oral loop diuretics and aldosterone antagonists (no dosage limitation)
* Because of the existence of excess body fluid retention, the congestive heart failure patient has at least one of these symptoms (the lower extremity edema, pulmonary congestion note 2), or jugular vein engorgement).
* 20-85 years of age (inclusive) at the time of signing the informed consent document.
* Gender: male or female.
* Inpatients or patient who would be hospitalized from one day before the observation period to the end of efficacy evaluation examination after the last dosing (from Day -4 to the end of efficacy evaluation examination after the last dosing).
* Patient who have signed the informed consent form.

Exclusion Criteria:

* Patients equipped with circulatory assistant device.
* Patients with any of following diseases, complications or symptoms:

  1. Suspected decreased blood volume
  2. Obstructive hypertrophic cardiomyopathy
  3. Severe aortic stenosis
  4. Hepatic coma
* Patients with history of acute myocardial infarction within 30 days prior to screening.
* Patients with diagnosed active myocarditis or amyloid cardiomyopathy.
* Patients with the following diseases, complications or symptoms:

  1. Poorly controlled diabetes with a fasting glucose more than 220 mg/dL (or 12.21 mmol/L)
  2. Anuria
  3. Dysuria caused by urethral stricture, calculus or tumor
* Patients with the following medical history of:

  1. Sustained ventricular tachycardia or ventricular fibrillation within 30 days prior to screening
  2. History of cerebrovascular accident within the past 30 days
  3. Past allergy or hypersensitive reactions to benzodiazepines (e.g. mozavaptan hydrochloride or benazepril hydrochloride)
* Obese patients whose body mass index (BMI = body weight (kg) / height (m)2 ) is more than 35.
* Patients with systolic pressure below 90 mmHg in supine position.
* Patients with any of the following abnormal laboratory test parameters:

  1. Total bilirubin > 2.5 times the upper limits of normal value
  2. Serum creatine > 2.5 times the upper limits of normal value
  3. Serum Na+ > 145 mmol/L (or higher than the upper limits of normal value)
  4. Serum K+ > 5.5 mmol/L
* Patients who unable to take medicine orally.
* Female patients who are pregnant, breast-feeding, at childbearing ages, or with pregnancy plan.
* Patients who participated in clinical trials of other medicine and took other study drugs within 30 days prior to sign the informed consent form.
* Patients who participated in the clinical trial of Tolvaptan and took Tolvaptan previously.
* Patients who have received approved Tolvaptan tablets (Trade name: Samsca) previously.
* Except for the above, patients who were unsuitable to participate in this trial in the investigator's opinion.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
body weight (change from baseline) | screening day, Day-3, Day-2, Day-1, Day1, Day2, Day3, Day4, Day5, Day6, Day7, Day8, Day(7+3)

SECONDARY OUTCOMES:
Body weight (percent change from baseline) | screening day, Day-3, Day-2, Day-1, Day1, Day2, Day3, Day4, Day5, Day6, Day7, Day8, Day(7+3)

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Jian, Principal Investigator — Fuwai Cardiovascular hospital
Locations (1):
- Zhejiang Hospital, Hangzhou, Zhejiang, China